CLINICAL TRIAL: NCT01297803
Title: Corneal Endothelial Cell Loss Following Trabeculectomy With mitomycin_c Application Before Versus After Sclera Flap Dissection
Brief Title: Comparison of Two Method Antimetabolites Application on Corneal Function in Trabeculectomy Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Shahin Yazdani, Ophthalmic Research center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8772
Record Dates: First submitted 2011-01-19; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2010-11

CONDITIONS: Glaucoma Patients Scheduled for Trabeculectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin_c application before sclera flap dissection (Active Comparator)
  Interventions: Drug: Mitomycin_c
- Mitomycin_c application after sclera flapdissection (Active Comparator)
  Interventions: Drug: Mitomycin_c

INTERVENTIONS:
Drug: Mitomycin_c — 0.02%.1,2,3,minutes match randomized in to two groups(before &after scleral flap dissection
  Arms: Mitomycin_c application before sclera flap dissection
Drug: Mitomycin_c — 0.02%.1,2,3,minutes match randomized in to two groups(before &after scleral flap dissection
  Arms: Mitomycin_c application after sclera flapdissection

SUMMARY:
Application of antimetabolite agents such as mitomycin_c has improved trabeculectomy results and better control of intraocular pressure complications such as corneal endothelial cell loss. However, Mitomycin_c can be applied remain a concern before or after sclera flap dissection. Mitomycin_c application after sclera flap dissection probably increases corneal endothelial cell loss. This study compares Mitomycin_c application two methods: before and after sclera flap dissection with regard to success rate and complication. patients on base of Mitomycin_c application time (1-2-3) minutes will be match randomise in to two groups( before and after sclera flap dissection) corneal. Endothelial cell density, polymorphism, polymegathism and intraocular pressure before and one month, three months, six months after surgery will measured.

ELIGIBILITY:
Inclusion Criteria:

* Age Range between 18 to 80 years old
* Trabeculectomy to JOAC, POAG, CACG, PXF, pigment dispersion syndrome.

Exclusion Criteria:

* Secondary glaucoma (active uveitis, NVG, specific syndromes such as axenfeld rieger, Iridocorneal Endothelial syndrome, aniridia, peters, etc).

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
corneal endothelial cell density | six month
  specular microscopy
corneal endothelial cell polymorphism | 6 months
  specular microscopy
corneal endothelial cell polymegathism | 6 months
  specular microscopy

SECONDARY OUTCOMES:
IOP (intra ocular pressure) | six months
  applanation tonometry

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Iran